CLINICAL TRIAL: NCT02986373
Title: A Phase 2 Single-Arm Open-Label Extension Study to Investigate Safety With Risankizumab in Psoriatic Arthritis Subjects Who Have Completed Week 24 Visit of Study M16-002 (1311.5)
Brief Title: A Study to Investigate Safety With Risankizumab in Psoriatic Arthritis Subjects Who Have Completed Week 24 Visit of Study M16-002 (NCT02719171)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-244; 2016-003113-94 (EudraCT Number)
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Results first posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Psoriatic Arthritis
Keywords: risankizumab; ABBV-066; BI655066
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Risankizumab (Experimental): Participants received open-label risankizumab 150 mg by subcutaneous injection at Weeks 0, 12, 24, and 36.
  Interventions: Biological: risankizumab

INTERVENTIONS:
Biological: risankizumab — Risankizumab administered by subcutaneous injection.
  Other Names: ABBV-066; BI 655066; SKYRIZI

SUMMARY:
This is an open-label extension (OLE) study to assess the efficacy, safety and tolerability of risankizumab in participants with psoriatic arthritis (PsA).

DETAILED DESCRIPTION:
Participants who had completed all doses of study drug and the Week 24 visit of M16-002 (NCT02719171; the lead-in study) were eligible to enroll in M16-244 (this study). Participants were allowed to either finish the Week 24 visit of the lead-in study and take the first dose of study drug for this study on the same day, or delay the start of this study up to 8 weeks if needed.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed all doses of study drug and Week 24 visit of the lead-in study.
* Women of childbearing potential who are sexually active, must agree to use at least one accepted method of contraception throughout the study, including 20 weeks after last dose of study drug is given.
* Women of childbearing potential must have a negative urine pregnancy test at Baseline (Week 0/V1).
* Participants must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any study specific procedures.
* Participant is judged to be in good health as determined by the Investigator.

Exclusion Criteria:

* Female participant who is pregnant, breastfeeding or is considering becoming pregnant during study participation, including 20 weeks after the last dose of study drug is given.
* Premature discontinuation of the study drug in the lead-in study for any reason.
* Use of a biologic treatment other than risankizumab since first dose of study drug in the lead-in study.
* Time elapsed is > 8 weeks since the Week 24 visit in the lead-in study.
* Active systemic infections during the last 2 weeks (exception: common cold) prior to the first dose, as assessed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-07-08 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Thakre N, D'Cunha R, Goebel A, Liu W, Pang Y, Suleiman AA. Population Pharmacokinetics and Exposure-Response Analyses for Risankizumab in Patients with Active Psoriatic Arthritis. Rheumatol Ther. 2022 Dec;9(6):1587-1603. doi: 10.1007/s40744-022-00495-0. Epub 2022 Sep 30. PMID 36178584
- [Derived] Mease PJ, Kellner H, Morita A, Kivitz AJ, Aslanyan S, Padula SJ, Topp AS, Eldred A, Behrens F, Papp KA. Long-Term Efficacy and Safety of Risankizumab in Patients with Active Psoriatic Arthritis: Results from a 76-Week Phase 2 Randomized Trial. Rheumatol Ther. 2022 Oct;9(5):1361-1375. doi: 10.1007/s40744-022-00474-5. Epub 2022 Aug 5. PMID 35931879
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had completed all doses of study drug and the Week 24 visit of M16-002 (NCT02719171; lead-in study) were eligible to enroll in M16-244 (this study).
Period: Overall Study
Arm/Group | Risankizumab
Started | 145
Completed | 106
Not Completed | 39
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 10
Not completed — Other | 24

BASELINE CHARACTERISTICS:
Population: Safety analysis set: consists of all participants who received at least 1 dose of study medication in Study M16-244.
Arm/Group | Risankizumab
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 138
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 119
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent events (TEAEs) are defined as an AE that began or worsened in severity after initiation of study drug and 20 weeks (140 days) after last dose. Abbreviations: NMSC=non-melanoma skin cancer
Time Frame: From the first dose of study drug in this study until 20 weeks after the last dose of study drug (up to 56 weeks).
Population: Safety Analysis Set: consists of all participants who have received at least 1 dose of study medication in Study M16-244 (this study).
Measure: Number; unit: participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 145
participants
  Any AE | 87
  Any AE at least possibly drug related | 22
  Any SAE at least possibly drug related | 1
  Any severe AE | 7
  Any SAE | 5
  Any AE leading to discontinuation of study drug | 5
  Any major adverse cardiac events (by adjudication) | 2
  Any Serious Infections Events | 2
  Any tuberculosis events | 2
  Any malignant tumor events | 1
  Any malignancies excluding NMSC events | 1

2. Secondary Outcome: Modified Total Sharp Score (mTSS): Change From Baseline (in the Lead-in Study) to Week 24 in the Lead-in Study
Description: The mTSS is a measure of change in joint health. X-rays of hands, wrists, and feet (including distal interphalangeal joints) were obtained at Week 24 and Week 48. Totals for hands and feet for erosion scores (range 0 to 320) and joint space narrowing scores (range 0 to 208) were calculated and added to obtain the mTSS (range = 0 [normal] to 528 [maximal disease]). An increase in mTSS from Baseline represents disease progression and/or joint worsening; no progression was defined as a change of ≤0.5. Baseline is defined as baseline in the lead-in study.
Time Frame: Baseline (Lead-in Study), Week 24 (Lead-in Study)
Population: Safety analysis set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 118
units on a scale | 0.12 [-0.16 to 0.40]

3. Secondary Outcome: mTSS: Change From Baseline (in the Lead-in Study) to Week 24
Description: as for outcome 2
Time Frame: Baseline (Lead-in Study), Week 24
Population: Safety analysis set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 118
units on a scale | 0.38 [0.06 to 0.71]

4. Secondary Outcome: mTSS: Change From Baseline (in the Lead-in Study) to Week 48
Description: as for outcome 2
Time Frame: Baseline (Lead-in Study), Week 48
Population: Safety analysis set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 102
units on a scale | 0.34 [-0.07 to 0.75]

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 0
Description: Response defined by ACR20 criteria (improvement from baseline in the lead-in study) at Week 0: ≥20% improvement in tender joint count; ≥20% improvement in swollen joint count; and ≥20% improvement in at least 3 out of the following 5 parameters: Patient's Assessment of Pain Intensity visual analog scale (VAS), Patient's Global Assessment of Disease Activity, Investigator's Global Assessment of Disease Activity, Health Assessment Questionnaire Disability Index (HAQ-DI), and acute phase reactant value (C-reactive protein). Baseline is defined as the last non missing pre-treatment observation prior to first dose in the lead-in study.
Time Frame: Week 0
Population: Safety analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 145
percentage of participants | 43.4 [35.2 to 51.9]

6. Secondary Outcome: Percentage of Participants Achieving ACR20 Response at Week 4
Description: Response defined by ACR20 criteria (improvement from baseline in the lead-in study) at Week 4: ≥20% improvement in tender joint count; ≥20% improvement in swollen joint count; and ≥20% improvement in at least 3 out of the following 5 parameters: Patient's Assessment of Pain Intensity VAS, Patient's Global Assessment of Disease Activity, Investigator's Global Assessment of Disease Activity, HAQ-DI, and acute phase reactant value (C-reactive protein). Baseline is defined as the last non missing pre-treatment observation prior to first dose in the lead-in study.
Time Frame: Week 4
Population: Safety analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 144
percentage of participants | 55.6 [47.1 to 63.8]

7. Secondary Outcome: Percentage of Participants Achieving ACR20 Response at Week 12
Description: Response defined by ACR20 criteria (improvement from baseline in the lead-in study) at Week 12: ≥20% improvement in tender joint count; ≥20% improvement in swollen joint count; and ≥20% improvement in at least 3 out of the following 5 parameters: Patient's Assessment of Pain Intensity VAS, Patient's Global Assessment of Disease Activity, Investigator's Global Assessment of Disease Activity, HAQ-DI, and acute phase reactant value (C-reactive protein). Baseline is defined as the last non missing pre-treatment observation prior to first dose in the lead-in study.
Time Frame: Week 12
Population: Safety analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 142
percentage of participants | 57.0 [48.5 to 65.3]

8. Secondary Outcome: Percentage of Participants Achieving ACR20 Response at Week 24
Description: Response defined by ACR20 criteria (improvement from baseline in the lead-in study) at Week 24: ≥20% improvement in tender joint count; ≥20% improvement in swollen joint count; and ≥20% improvement in at least 3 out of the following 5 parameters: Patient's Assessment of Pain Intensity VAS, Patient's Global Assessment of Disease Activity, Investigator's Global Assessment of Disease Activity, HAQ-DI, and acute phase reactant value (C-reactive protein). Baseline is defined as the last non missing pre-treatment observation prior to first dose in the lead-in study.
Time Frame: Week 24
Population: Safety analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 134
percentage of participants | 62.7 [53.9 to 70.9]

9. Secondary Outcome: Percentage of Participants Achieving ACR20 Response at Week 36
Description: Response defined by ACR20 criteria (improvement from baseline in the lead-in study) at Week 36: ≥20% improvement in tender joint count; ≥20% improvement in swollen joint count; and ≥20% improvement in at least 3 out of the following 5 parameters: Patient's Assessment of Pain Intensity VAS, Patient's Global Assessment of Disease Activity, Investigator's Global Assessment of Disease Activity, HAQ-DI, and acute phase reactant value (C-reactive protein). Baseline is defined as the last non missing pre-treatment observation prior to first dose in the lead-in study.
Time Frame: Week 36
Population: Safety analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 115
percentage of participants | 68.7 [59.4 to 77.0]

10. Secondary Outcome: Percentage of Participants Achieving ACR20 Response at Week 48
Description: Response defined by ACR20 criteria (improvement from baseline in the lead-in study) at Week 48: ≥20% improvement in tender joint count; ≥20% improvement in swollen joint count; and ≥20% improvement in at least 3 out of the following 5 parameters: Patient's Assessment of Pain Intensity VAS, Patient's Global Assessment of Disease Activity, Investigator's Global Assessment of Disease Activity, HAQ-DI, and acute phase reactant value (C-reactive protein). Baseline is defined as the last non missing pre-treatment observation prior to first dose in the lead-in study.
Time Frame: Week 48
Population: Safety analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 109
percentage of participants | 69.7 [60.2 to 78.2]

11. Secondary Outcome: Percentage of Participants Achieving ACR20 Response at Week 52
Description: Response defined by ACR20 criteria (improvement from baseline in the lead-in study) at Week 52: ≥20% improvement in tender joint count; ≥20% improvement in swollen joint count; and ≥20% improvement in at least 3 out of the following 5 parameters: Patient's Assessment of Pain Intensity VAS, Patient's Global Assessment of Disease Activity, Investigator's Global Assessment of Disease Activity, HAQ-DI, and acute phase reactant value (C-reactive protein). Baseline is defined as the last non missing pre-treatment observation prior to first dose in the lead-in study.
Time Frame: Week 52
Population: Safety analysis set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risankizumab
Number analyzed (Participants) | 101
percentage of participants | 75.2 [65.7 to 83.3]

12. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI): Change From Baseline (in the Lead-in Study) to Week 0
Description: The HAQ-DI is a patient-reported questionnaire specific for rheumatoid arthritis that consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 very severe, high-dependency disability. HAQ remission indicating normal physical function is defined by HAQ-DI score of < 0.5. Negative change from Baseline indicates improvement. Baseline is defined as baseline in the lead-in study.
Time Frame: Baseline (Lead-in Study), Week 0
Population: Safety analysis set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 143
units on a scale | -0.176 [-0.249 to -0.102]

13. Secondary Outcome: HAQ-DI: Change From Baseline (in the Lead-in Study) to Week 4
Description: as for outcome 12
Time Frame: Baseline (Lead-in Study), Week 4
Population: Safety analysis set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 143
units on a scale | -0.258 [-0.332 to -0.183]

14. Secondary Outcome: HAQ-DI: Change From Baseline (in the Lead-in Study) to Week 12
Description: as for outcome 12
Time Frame: Baseline (Lead-in Study), Week 12
Population: Safety analysis set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 140
units on a scale | -0.261 [-0.336 to -0.186]

15. Secondary Outcome: HAQ-DI: Change From Baseline (in the Lead-in Study) to Week 24
Description: as for outcome 12
Time Frame: Baseline (Lead-in Study), Week 24
Population: Safety analysis set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 133
units on a scale | -0.296 [-0.374 to -0.217]

16. Secondary Outcome: HAQ-DI: Change From Baseline (in the Lead-in Study) to Week 36
Description: as for outcome 12
Time Frame: Baseline (Lead-in Study), Week 36
Population: Safety analysis set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 114
units on a scale | -0.294 [-0.384 to -0.204]

17. Secondary Outcome: HAQ-DI: Change From Baseline (in the Lead-in Study) to Week 48
Description: as for outcome 12
Time Frame: Baseline (Lead-in Study), Week 48
Population: Safety analysis set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 107
units on a scale | -0.298 [-0.381 to -0.215]

18. Secondary Outcome: HAQ-DI: Change From Baseline (in the Lead-in Study) to Week 52
Description: as for outcome 12
Time Frame: Baseline (Lead-in Study), Week 52
Population: Safety analysis set.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 99
units on a scale | -0.318 [-0.405 to -0.231]

19. Secondary Outcome: Short Form Health Survey 36 (SF-36) Physical Component Summary (PCS) Score: Change From Baseline (in the Lead-in Study) to Week 0
Description: The SF-36 Health determined participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 comprise the physical component of the SF-36. Scores on each item were summed and averaged (range = 0-100); a positive change from Baseline indicates improvement. Baseline is defined as baseline in the lead-in study.
Time Frame: Baseline (Lead-in Study), Week 0
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 144
units on a scale | 2.11 [0.89 to 3.34]

20. Secondary Outcome: SF-36 PCS Score: Change From Baseline (in the Lead-in Study) to Week 4
Description: as for outcome 19
Time Frame: Baseline (Lead-in Study), Week 4
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 143
units on a scale | 3.63 [2.41 to 4.85]

21. Secondary Outcome: SF-36 PCS Score: Change From Baseline (in the Lead-in Study) to Week 12
Description: as for outcome 19
Time Frame: Baseline (Lead-in Study), Week 12
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 140
units on a scale | 3.63 [2.32 to 4.94]

22. Secondary Outcome: SF-36 PCS Score: Change From Baseline (in the Lead-in Study) to Week 24
Description: as for outcome 19
Time Frame: Baseline (Lead-in Study), Week 24
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 134
units on a scale | 3.76 [2.50 to 5.02]

23. Secondary Outcome: SF-36 PCS Score: Change From Baseline (in the Lead-in Study) to Week 36
Description: as for outcome 19
Time Frame: Baseline (Lead-in Study), Week 36
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 115
units on a scale | 4.27 [2.97 to 5.57]

24. Secondary Outcome: SF-36 PCS Score: Change From Baseline (in the Lead-in Study) to Week 48
Description: as for outcome 19
Time Frame: Baseline (Lead-in Study), Week 48
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 108
units on a scale | 5.08 [3.66 to 6.50]

25. Secondary Outcome: SF-36 PCS Score: Change From Baseline (in the Lead-in Study) to Week 52
Description: as for outcome 19
Time Frame: Baseline (Lead-in Study), Week 52
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 100
units on a scale | 4.47 [3.11 to 5.84]

26. Secondary Outcome: SF-36 Mental Component Summary (MCS) Score: Change From Baseline (in the Lead-in Study) to Week 0
Description: The SF-36 determined participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 5-8 comprise the mental component of the SF-36. Scores on each item were summed and averaged (range = 0-100); a positive change from Baseline indicates improvement. Baseline is defined as baseline in the lead-in study.
Time Frame: Baseline (Lead-in Study), Week 0
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 144
units on a scale | 0.86 [-0.64 to 2.35]

27. Secondary Outcome: SF-36 MCS Score: Change From Baseline (in the Lead-in Study) to Week 4
Description: as for outcome 26
Time Frame: Baseline (Lead-in Study), Week 4
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 143
units on a scale | 2.79 [1.27 to 4.31]

28. Secondary Outcome: SF-36 MCS Score: Change From Baseline (in the Lead-in Study) to Week 12
Description: as for outcome 26
Time Frame: Baseline (Lead-in Study), Week 12
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 140
units on a scale | 2.22 [0.49 to 3.96]

29. Secondary Outcome: SF-36 MCS Score: Change From Baseline (in the Lead-in Study) to Week 24
Description: as for outcome 26
Time Frame: Baseline (Lead-in Study), Week 24
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 134
units on a scale | 4.08 [2.39 to 5.77]

30. Secondary Outcome: SF-36 MCS Score: Change From Baseline (in the Lead-in Study) to Week 36
Description: as for outcome 26
Time Frame: Baseline (Lead-in Study), Week 36
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 115
units on a scale | 3.44 [1.60 to 5.28]

31. Secondary Outcome: SF-36 MCS Score: Change From Baseline (in the Lead-in Study) to Week 48
Description: as for outcome 26
Time Frame: Baseline (Lead-in Study), Week 48
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 108
units on a scale | 3.36 [1.40 to 5.31]

32. Secondary Outcome: SF-36 MCS Score: Change From Baseline (in the Lead-in Study) to Week 52
Description: as for outcome 26
Time Frame: Baseline (Lead-in Study), Week 52
Population: Safety analysis set.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Risankizumab
Number analyzed (Participants) | 100
units on a scale | 4.33 [2.56 to 6.10]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug in this study until 20 weeks after the last dose of study drug (up to 56 weeks).
Arm/Group | Risankizumab
All-Cause Mortality (participants affected / at risk) | 0/145
Serious Adverse Events (participants affected / at risk) | 5/145
Other Adverse Events (participants affected / at risk) | 16/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab (N=145)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 1 (1)
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 1 (1)
PNEUMONIA HAEMOPHILUS (Infections and infestations) | 1 (1)
PNEUMONIA PSEUDOMONAL (Infections and infestations) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1)
UROSEPSIS (Infections and infestations) | 1 (1)
GLOMERULAR FILTRATION RATE ABNORMAL (Investigations) | 1 (1)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risankizumab (N=145)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 16 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT02986373/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT02986373/SAP_001.pdf